CLINICAL TRIAL: NCT07286396
Title: Non-invasive Intracranial Pressure Monitoring in Brain Tumor Patients: A Prospective Observational Study of Optic Nerve Sheath Diameter Dynamics
Brief Title: Non-invasive Intracranial Pressure Monitoring in Brain Tumor Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: ICP measurement
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Brain Neoplasm; Intracranial Pressure Increase
MeSH Terms: conditions — Brain Neoplasms; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ocular Sonography — The examination will employ an ultrasound machine with a linear probe. Patients will be positioned supine with their heads elevated at a 20-30° angle. They will be instructed to keep their eyes closed in a neutral position while suppressing voluntary eye movement.The transducer will be gently placed on the gel in the temporal region of the eyelid to avoid exerting pressure on the eye. Optic nerve sheath diameter will be measured 3 mm posterior to the optic nerve's tip, with electronic calipers used to measure the values. ONSD will be defined as the distance within the dura mater, and ETD will be measured across the maximal transverse diameter of the eyeball, from one side of the retina behind the lens to the other. Measurements will be taken in both coronal and sagittal planes by positioning the probe perpendicular (90°) to the coronal plane, ensuring optimal alignment of the optic nerve with the probe.

SUMMARY:
This research protocol focuses on the pre- and post-operative evaluation of ICP using non-invasive methods, particularly in the context of surgery for brain tumor removal. By utilizing ocular ultrasound to measure ONSD and ONSD/ETD ratios, this study hypothesizes that the utility of these parameters in monitoring ICP pre- and post-operative periods could be effective.

DETAILED DESCRIPTION:
This research protocol focuses on the pre- and post-operative evaluation of ICP using non-invasive methods, particularly in the context of brain tumor resection surgery. By utilizing ocular ultrasound to measure ONSD and ONSD/ETD ratios, this study hypothesizes that the utility of these parameters in monitoring ICP pre- and post-operative periods could be effective.

This study aims to evaluate the effectiveness of the ONSD and the ONSD/ETD ratio using ultrasound as a non-invasive method for measuring intracranial pressure pre- and post-operatively in brain tumor patients.

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (>21 years) undergoing brain tumor resection surgery.

  * Preoperative imaging-confirmed diagnosis of the tumor.
  * American Society of Anesthesiologists (ASA) physical status II to IV
  * Consent to participate in the study.

Exclusion Criteria:

* • Preexisting ocular conditions affecting the optic nerve or globe integrity, such as glaucoma, thyroid-associated ophthalmopathy, or other optic nerve diseases.

  * Combined ocular and optic nerve injuries at admission.
  * History of cranial trauma, prior neurosurgery, or lumbar puncture performed within 2 weeks before the measurement of optic nerve sheath diameter (ONSD).
  * History of subarachnoid hemorrhage (SAH).
  * Serious complications that could affect life expectancy, such as hematological disorders or malignancies.
  * Refusal to participate or withdrawal of consent at any stage.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study that will be conducted on 60 adult patients aged more than 21 years with ASA physical status II or IV. These patients will be admitted for brain tumor resection surgery at Tanta University Hospitals undergoing brain tumor resection surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
optic nerve sheath diameter dynamics | before (in the preoperative holding area) and after the surgery (immediate, 1,2, 4, 6, and 12 hr in ICU).
  the measuremnt of optic nerve sheath diameter and optic nerve sheath diameter to transverse eyeball diamter ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided